CLINICAL TRIAL: NCT05682170
Title: A Phase 1/2 Dose Escalation Study of the BCL-2 Inhibitor ZN-d5 and the WEE1 Inhibitor ZN-c3 in Subjects With Acute Myeloid Leukemia
Brief Title: Study of the ZN-d5 and ZN-c3 in Subjects With Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: K-Group Alpha, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZN-d5-004C
Record Dates: First submitted 2022-12-19; First posted 2023-01-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: BCL-2 Inhibitors; Wee1 Inhibitors; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acute Myeloid Leukemia (Experimental): Phase 1: Dose Escalation- c3 monotherapy and d5+c3 combination
  Phase 2: Dose Expansion
  Interventions: Drug: ZN-d5 ZN-c3; Drug: ZN-c3

INTERVENTIONS:
Drug: ZN-d5 ZN-c3 — Oral agent
  Other Names: Study Drug
Drug: ZN-c3 — Oral agent
  Other Names: Study Drug

SUMMARY:
A Phase 1/2 dose escalation study of BCL-2 Inhibitor ZN-d5 and the Wee1 Inhibitor ZN-c3 in Subjects with Acute Myeloid Leukemia (AML).

DETAILED DESCRIPTION:
This is an open-label multicenter Phase 1/2 dose escalation study, evaluating the safety, tolerability, clinical activity, pharmacokinetics and pharmacodynamics of the novel BCL-2 inhibitor ZN-d5 and Wee1 inhibitor ZN-c3 in subjects with AML.

ELIGIBILITY:
Inclusion Criteria:

* Adults with AML (including secondary or therapy-related), relapsed from or refractory to one or more prior lines of therapy, which may include venetoclax except in Expansion Cohort A
* ECOG performance status score ≤2.
* Projected life expectancy of at least 12 weeks.
* Estimated glomerular filtration rate ≥60 mL/min
* Women of childbearing potential must not be pregnant and must use effective birth control during the study and for 6 months after the last dose of study drugs.
* Men must agree to use a condom when having intercourse during the study and for 3 months after the last dose of study drugs.

Exclusion Criteria:

* Known active CNS involvement
* Diagnosis of acute promyelocytic leukemia.
* Peripheral blast count of >25 × 109/L (cytoreduction permitted).
* Adequate washout from prior therapy including hematopoietic stem cell transplant and recovery from prior treatment-related toxicities to Grade 2 or lower
* Significant cardiovascular disease
* Corrected QT interval (QTc) of >480 msec
* Active hepatitis B or hepatitis C infection
* Concurrent treatment with strong CYP3A inhibitors or strong or moderate CYP3A inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Observed dose limiting toxicities | At the end of Cycle 1 (each cycle is 28 days)
  Observed Dose Limiting Toxicities (DLTs) in DLT evaluable subjects.
Incidence, severity, and relatedness of adverse events( AEs) | Through study completion, typically < 12 months

SECONDARY OUTCOMES:
1. To investigate the plasma PK of ZN-c3 when given as monotherapy - Maximum Plasma Concentration | Through study completion, typically <12 months
  The maximum plasma concentration (Cmax) of ZN-c3 (and its potential metabolites, as applicable) will be determined
2. To investigate the plasma PK of ZN-c3 when given as monotherapy - Area under the plasma concentration-time curve from 0 to 24h | Through study completion, typically < 12 months
  Area under the plasma concentration-time curve from 0 to 24h [AUC0-24h] of ZN-c3 (and its potential metabolites, as applicable) will be determined
5. To investigate the plasma PK of ZN-c3 and ZN-d5 when given in combination - Maximum Plasma Concentration | Through study completion, typically < 12 months
  The maximum plasma concentration (Cmax) of ZN-c3 (and its potential metabolites, as applicable) and ZN-d5 (and its potential metabolites, as applicable) will be determined
6. To investigate the plasma PK of ZN-c3 and ZN-d5 when given in combination - Area under the plasma concentration-time curve from 0 to 24h | Through study completion, typically < 12 months
  Area under the plasma concentration-time curve from 0 to 24h [AUC0-24h] of ZN-c3 (and its potential metabolites, as applicable) and ZN-d5 (and its potential metabolites, as applicable) will be determined
Rate and duration or remission according to the European LeukemiaNet 2017 criteria | Through study completion, typically < 12 months

CONTACTS AND LOCATIONS:
Overall Officials: K-Group Alpha, Inc. a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc., Study Director — K-Group Alpha
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Albert Einstein College of Medicine - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Tristar Bone Marrow Transplant, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No